CLINICAL TRIAL: NCT06588894
Title: Relationship Between Motor Imagery Ability, Body Awareness and Cognitive Functions in Individuals With Type 2 Diabetes Mellitus
Brief Title: Investigation of Motor Imagery Ability, Body Awareness and Cognitive Functions in Type 2 Diabetes Mellitus
Status: Recruiting | Type: Observational
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Principal Investigator, Ismail Okur, Assist. Prof., Kutahya Health Sciences University
Other Study IDs: 2024/03-26
Record Dates: First submitted 2024-09-05; First posted 2024-09-19 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Type 2 Diabetes Mellitus (T2DM); Cognitive Function; Motor İmagery Ability
Keywords: cognitive functions; motor imagery ability; type 2 diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Surveys and Questionnaires; Restraint, Physical; Neuropsychological Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Type 2 Diabetes Mellitus: 18-65 years old with type 2 DM for at least 5 years
  Interventions: Behavioral: Questionnaire and Physical Exam; Behavioral: Motor Imagery Ability

INTERVENTIONS:
Behavioral: Questionnaire and Physical Exam — Individuals motor imagery skills will be assessed using a mental chronometer and mental rotation, body awareness will be assessed using the Body Awareness Questionnaire, and cognitive functions will be assessed using the Montreal Cognitive Assessment questionnaire.
  Other Names: Cognitive Function; Motor imagery Ability; Body Awareness
Behavioral: Motor Imagery Ability — Individuals motor imagery skills will be assessed using a mental stopwatch and mental rotation, body awareness will be assessed using the Body Awareness Questionnaire, and cognitive functions will be assessed using theMontreal Cognitive Assessment questionnaire.
  Other Names: Cognitive Function; Body Awareness

SUMMARY:
The aim of this study is to examine the relationship between motor imagery skills, body awareness and cognitive functions in individuals with Type 2 Diabetes mellitus.

DETAILED DESCRIPTION:
Motor imagery can be defined as a voluntary action simulation process that involves focusing intently on the cognitive components of motor tasks. In the literature, motor imagery is seen as a window opening to cognitive motor processes and especially motor control. Motor imagery is negatively affected in many diseases that affect the brain and brain functions, such as stroke, Parkinson, and multiple sclerosis, and motor imagery is frequently used in the rehabilitation of these diseases. Poor glycemic control in Type 2 Diabetes mellitus leads to deterioration in brain and cognitive functions. However, no study has been found on the effects of these disorders seen in Type 2 Diabetes mellitus on MI skills. Motor imagery is a mental practice that is becoming widespread in many areas. However, before considering using Motor imagery-based exercises as a therapy tool for patients, it is important to consider the extent to which patients cognitive impairments are related to their ability to form accurate motor images. For example, studies have found that patients with the lack of body awareness may not be able to produce kinesthetic images of motor movements.

Body awareness is the tendency to pay attention to internal bodily sensations and stimuli and includes the cognitive, emotional, and perceptual abilities that constitute the person general self-awareness. Chronic diseases such as Type 2 Diabetes mellitus affect body awareness and image. Body awareness has been found to be associated with clinical parameters related to diabetes, such as fasting blood sugar and HbA1c levels and duration of diabetes in patients with Type 2 Diabetes mellitus. Changes in body awareness may disrupt the patient self-perception, leading to a poor clinical picture and a poor course of chronic diseases. Therefore, it is important to evaluate possible changes in internal body perception.

To our knowledge, no study has been found in the literature examining the relationship between motor imagery skills of individuals with type 2 diabetes mellitus and body awareness and cognitive functions. The existence of this relationship may guide the use of motor imagery as a treatment method in individuals with Type 2 Diabetes mellitus whose body awareness and cognitive functions are impaired.

Individuals who meet the inclusion criteria will be asked to sign an informed consent form. Then, demographic data of the individuals will be collected using a demographic data form. Individuals; motor imagery skills will be assessed using a mental stopwatch and mental rotation, body awareness will be assessed using the Body Awareness Questionnaire, and cognitive functions will be assessed using the Montreal Cognitive Assessment questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Being a type 2 DM patient between the ages of 18-65 for at least 5 years,
* Being willing to participate in the study,
* Not having any vision, hearing or speech problems that would prevent the tests from being performed.

Exclusion Criteria:

* Having previous experience with Motor Imagery techniques or training,
* Having any orthopedic problems that prevent walking,
* Having a history of neurological disease,
* People who are receiving any medication that affects the central nervous system will not be included in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals aged 18-65 who have had type 2 DM for at least 5 years
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-10-14 (Actual); Primary Completion 2025-11-14 (Estimated); Study Completion 2025-12-10 (Estimated)

PRIMARY OUTCOMES:
Mental Chronometer | 10 minutes
  Mental chronometry provides information about the temporal relationship between real and simulated movements. As part of this assessment, participants will be administered the Nine-Hole Wooden Peg Test. In the study, the patient will be asked to place wooden sticks in the box one by one into the holes on the board as quickly as possible with their dominant hand. They will then be asked to place the sticks back into the box one by one. The total duration of the test will be determined by a chronometer. After the materials are removed from the field of vision, they will be asked to perform this carrying activity using the imagery method and the elapsed time will again be recorded by a chronometer. Motor imagery trials will begin with a countdown of "3-2-1-Start" and will end when participants indicate that they have finished placing by saying "stop".
Mental Rotation | 10 minutes
  Mental rotation provides information about the accuracy of imagined movements. Mental rotation will be evaluated as a hand lateralization task, which is choosing which side the hand belongs to. The test will be applied using the Recognize App Recognize Hand software (Neuro Orthopedic Institute, Adelaide, Australia). Two data will be obtained by performing the test. The first is the percentage of correct responses that are capable of understanding whether the hand images shown belong to the right or the left, and the second is the reaction times of the individuals while performing the task. The "Vanilla" mode will be used for mental rotation ability in the study. This mode consists of images of real human hands in different postures/positions. The patient is given 5 seconds for each hand image and is expected to indicate whether the hand in the image is right or left from the buttons below during this time.
Body Awareness | 10 minutes
  Individuals; body awareness will be measured with the Body Awareness Questionnaire. The Body Awareness Questionnaire consists of 18 questions. Participants will be asked to score each statement between 1 (1: Not true for me at all) and 7 (7: Completely true for me), and the total score is obtained by adding the scores given for each statement. The total score takes a value between 18 and 126. The higher the total score, the better the body awareness.
Cognitive Function | 20 minutes
  Cognitive functions will be assessed with the Montreal Cognitive Assessment (MOCA) questionnaire. MOCA is a screening test that assesses attention and concentration, executive functions, memory, language, visual-spatial abilities, abstract thinking, calculation, and orientation. The total score on the MOCA test ranges from 0 to 30. The cutoff for a normal MOCA score is 26.

CONTACTS AND LOCATIONS:
Overall Officials: İsmail Okur, PhD, Principal Investigator — Kutahya Health Sciences University
Locations (1):
- Kutahya Health Sciences University, Kütahya, Central, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No